CLINICAL TRIAL: NCT00796848
Title: Reversal of Hypoglycemia Unawareness Using Continuous Glucose Monitoring
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: withdrawn because the research efforts at that time followed another path
Sponsor: Stanford University (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Bruce A. Buckingham, Principle Investigator, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SU-10172008-1323; Stanford eprotocol #14728 (Other: Stanford IRB)
Record Dates: First submitted 2008-10-23; First posted 2008-11-24 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Navigator Continuous Glucose Monitor

SUMMARY:
The purpose of doing this study is to see if continuous glucose monitoring can help people with type 1 diabetes who are sometimes unable to feel if they have a low blood glucose reading. For this study we will be using the Navigator Continuous Glucose Monitor. We think that your body may not have enough of a certain hormone that usually helps people know when they are going low. If you can keep from going low, we think there will be enough of that hormone to help you recognize the symptoms of a low before it happens.

DETAILED DESCRIPTION:
To enroll in this study you must be between the ages of 7 and 20, have type 1 diabetes, and experience at least two episodes of low blood glucose readings weekly that you do not feel. Up to 25 subjects will be enrolled at Stanford and another 25 at the Barbara Davis Center in Colorado. The study will last approximately 8 months for each participant.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 7 to 20 years old
2. Have been diagnosed with type 1 diabetes for at least 1 year
3. Report 2 or more episodes per week of asymptomatic hypoglycemia as determined by completion of the Hypoglycemia Awareness Questionnaire (HAQ) or as determined by Investigator
4. HbA1c level < 10%
5. Internet access for downloading continuous glucose monitoring (CGM), access to a compatible computer (Windows Vista is not compatible for downloading.)
6. For females, you are not intending to become pregnant during the study
7. No expectation that you will be moving out of the area for the duration of the study

Exclusion Criteria:

1. The presence of a significant medical disorder (including epilepsy, or any cause of seizures other than hypoglycemia) that in the judgment of the Investigator will affect the wearing of the sensors or the completion of any aspect of the protocol
2. Treatment with systemic or inhaled corticosteroids in the last six months
3. Inpatient psychiatric treatment in the past six months for you or your primary caregiver
4. Current use of oral/inhaled glucocorticoids or other medications, which in the judgment of the Investigator would be a contraindication to participation in the study
5. Having two or more severe hypoglycemia episodes (seizure or loss of consciousness) in the six months prior to enrollment
6. Having a severe hypoglycemic episode in the 30 days prior to enrollment

Ages: 7 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of continuous glucose monitoring in the reduction of hypoglycemia unawareness.

SECONDARY OUTCOMES:
To assess the levels of epinephrine production in youth diagnosed with hypoglycemia unawareness with and without continuous glucose monitor wear.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A. Buckingham, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- See also: Stanford Pediatric Endocrinology Department website — http://dped.stanford.edu/